CLINICAL TRIAL: NCT02354534
Title: A Phase I Study of Intravaginally Administered Artesunate In Women With High Grade Cervical Intraepithelial Neoplasia (CIN2/3)
Brief Title: Intravaginal Artesunate for the Treatment of HPV+ High Grade Cervical Intraepithelial Neoplasia (CIN2/3)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Frantz Viral Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1498; IRB00045376 (Other: JHM IRB)
Record Dates: First submitted 2015-01-13; First posted 2015-02-03 (Estimated); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-03

CONDITIONS: Cervical Intraepithelial Neoplasia Grade 2/3; High-risk HPV (Any Strain)
Keywords: cervical dysplasia; HPV; Treatment; preinvasive; cervix; vaginal suppository; Cornelia Trimble; abnormal pap; CIN
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 50 mg Artesunate suppositories, 1 cycle (Experimental): Subjects enrolled in this cohort will receive 1 five day cycle of Artesunate suppositories prior to therapeutic resection of their lesion (if clinically indicated).
  Interventions: Drug: Artesunate Suppositories
- 200 mg Artesunate suppositories, 1 cycle (Experimental): Subjects enrolled in this cohort will receive 1 five day cycle of Artesunate suppositories prior to therapeutic resection of their lesion (if clinically indicated).
  Interventions: Drug: Artesunate Suppositories
- 200 mg Artesunate suppositories,2 cycles (Experimental): Subjects enrolled in this cohort will receive 2 five day cycles of Artesunate suppositories prior to therapeutic resection of their lesion (if clinically indicated).
  Interventions: Drug: Artesunate Suppositories
- 200 mg Artesunate suppositories,3 cycles (Experimental): Subjects enrolled in this cohort will receive 3 five day cycles of Artesunate suppositories prior to therapeutic resection of their lesion (if clinically indicated).
  Interventions: Drug: Artesunate Suppositories

INTERVENTIONS:
Drug: Artesunate Suppositories

SUMMARY:
This phase I research protocol is designed to assess immunogenicity and clinical endpoints in patients with human papillomavirus (HPV) 16 cervical intraepithelial neoplasia (CIN)2/3. The protocol tests the use of artesunate in suppository formulation applied intravaginally in patients with cervical dysplasia (CIN2/3).

The primary endpoint is to determine and evaluate the safety, tolerability, and feasibility of intravaginal administration of artesunate in health women with CIN2/3.

DETAILED DESCRIPTION:
Phase I open-label dose escalation study of intravaginal artesunate, formulated in suppositories, in adult females with biopsy-confirmed CIN2/3. Thirty (30) subjects will undergo up to a total of three cycles of intravaginal artesunate. The first cycle will be initiated on Day 0, the second at Week 4, and the third and final cycle at week 8.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Capable of informed consent
* HPV-positive by DNA test
* Histologically confirmed CIN 2, CIN 3, or CIN 2/3
* Body weight ≥ 50 kg
* Immune competent

Exclusion Criteria:

* Pregnant and nursing women
* HIV seropositive
* Active autoimmune disease
* Taking immunosuppressive medication
* Evidence of concurrent adenocarcinoma in situ
* Concurrent malignancy except for nonmelanoma skin lesions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia L Trimble, MD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Johns Hopkins Outpatient Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Greater Baltimore Medical Center, Towson, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 50 mg Artesunate Suppositories, 1 Cycle; 200 mg Artesunate Suppositories, 1 Cycle: Subjects enrolled in this cohort will receive 1 five day cycle of Artesunate suppositories prior to therapeutic resection of their lesion (if clinically indicated).
  Artesunate Suppositories
- 200 mg Artesunate Suppositories,2 Cycles: Subjects enrolled in this cohort will receive 2 five day cycles of Artesunate suppositories prior to therapeutic resection of their lesion (if clinically indicated).
  Artesunate Suppositories
- 200 mg Artesunate Suppositories,3 Cycles: Subjects enrolled in this cohort will receive 3 five day cycles of Artesunate suppositories prior to therapeutic resection of their lesion (if clinically indicated).
  Artesunate Suppositories
Period: Overall Study
Arm/Group | 50 mg Artesunate Suppositories, 1 Cycle | 200 mg Artesunate Suppositories, 1 Cycle | 200 mg Artesunate Suppositories,2 Cycles | 200 mg Artesunate Suppositories,3 Cycles
Started | 3 | 9 | 10 | 8
Completed | 3 | 9 | 9 | 8
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 50 mg Artesunate Suppositories, 1 Cycle | 200 mg Artesunate Suppositories, 1 Cycle | 200 mg Artesunate Suppositories,2 Cycles | 200 mg Artesunate Suppositories,3 Cycles | Total
Number analyzed (Participants) | 3 | 9 | 10 | 8 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 9 | 10 | 8 | 30
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 10 | 8 | 30
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 0 | 2 | 1 | 2 | 5
  White | 3 | 7 | 7 | 4 | 21
  Asian | 0 | 0 | 2 | 1 | 3
  Hispanic | 0 | 1 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 9 | 10 | 8 | 30
Type of HPV at baseline [Count of Participants; unit: Participants]
  HPV16 only | 0 | 3 | 1 | 4 | 8
  HPV16 and other genotypes | 0 | 2 | 2 | 0 | 4
  Non-16 HPV genotypes | 3 | 4 | 7 | 4 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events
Description: Number of participants with serious adverse events or dose limiting toxicities related to the study intervention assessed using Common Terminology Criteria for Adverse Events (CTCAE) 4.0 criteria.
Time Frame: 41 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg Artesunate Suppositories, 1 Cycle | 200 mg Artesunate Suppositories, 1 Cycle | 200 mg Artesunate Suppositories,2 Cycles | 200 mg Artesunate Suppositories,3 Cycles
Number analyzed (Participants) | 3 | 9 | 10 | 8
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Viral Clearance of HPV
Description: Number of participants whose human papillomavirus (HPV) genotypes present at study entry become undetectable without surgical intervention. HPV genotyping detects strains of HPV present at each timepoint. For this outcome, we evaluated whether strains of HPV detected at study entry became undetectable during the study participation.
Time Frame: 41 weeks
Population: Subjects enrolled in the study who received at least one dose of the investigational drug, and on whom we have outcomes data. 2 participants did not have data collected for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg Artesunate Suppositories, 1 Cycle | 200 mg Artesunate Suppositories, 1 Cycle | 200 mg Artesunate Suppositories,2 Cycles | 200 mg Artesunate Suppositories,3 Cycles
Number analyzed (Participants) | 3 | 9 | 8 | 8
Participants | 1 | 3 | 4 | 1

3. Secondary Outcome: Histologic Regression of CIN2/3
Description: Number of participants who had histologic regression from cervical intraepithelial neoplasia (CIN) 2/3 to CIN 1 or less, as assessed by colposcopically-directed biopsies. Histologic regression is defined as disappearance of the high grade lesion (CIN2/3) without surgical intervention.
Time Frame: 41 weeks
Population: All participants who received at least one dose of the interventional drug and on whom we have outcomes data. 2 participants did not have data collected for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | 50 mg Artesunate Suppositories, 1 Cycle | 200 mg Artesunate Suppositories, 1 Cycle | 200 mg Artesunate Suppositories,2 Cycles | 200 mg Artesunate Suppositories,3 Cycles
Number analyzed (Participants) | 3 | 9 | 8 | 8
Participants | 2 | 7 | 5 | 5

ADVERSE EVENTS:
Time Frame: 41 weeks
Description: All adverse events reported by study participants from the time of study drug administration through 30 days after the final treatment, whether or not they are related to the study intervention.
  Participants filled out a symptom diary for each treatment cycle completed. Adverse events were also documented and assessed for causality by the study investigators at each study visit.
Arm/Group | 50 mg Artesunate Suppositories, 1 Cycle | 200 mg Artesunate Suppositories, 1 Cycle | 200 mg Artesunate Suppositories,2 Cycles | 200 mg Artesunate Suppositories,3 Cycles
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/9 | 0/10 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/9 | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 2/3 | 9/9 | 8/10 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 mg Artesunate Suppositories, 1 Cycle (N=3) | 200 mg Artesunate Suppositories, 1 Cycle (N=9) | 200 mg Artesunate Suppositories,2 Cycles (N=10) | 200 mg Artesunate Suppositories,3 Cycles (N=8)
Bloating (Gastrointestinal disorders) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) — Ringing in the ear
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Loss in appetite
Salivary duct inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Change in taste
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 2 (2) | 4 (4) | 1 (2) — bacterial or yeast infections
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vaginal twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 2 (6) | 3 (5) | 3 (3) — sensation of movement, unsteadiness
Headache (Nervous system disorders) | 1 (2) | 5 (9) | 3 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — painful urination
Uterine cramping (Reproductive system and breast disorders) | 2 (5) | 1 (3) | 1 (1) | 2 (2)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 1 (4) | 3 (4)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (1) — pruritus due to dryness
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) — light spotting
vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
vaginal pain/burning (Reproductive system and breast disorders) | 0 (0) | 4 (5) | 4 (4) | 4 (7)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — eczema
pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — body itching
Vaginal pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 5 (5) | 6 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT02354534/Prot_SAP_000.pdf